CLINICAL TRIAL: NCT05221047
Title: Translation and Validation Study of the Urdu Version of the Knee Outcome Survey-Activities of Daily Living Scale in Patients With Knee Osteoarthritis
Brief Title: A Reliability and Validity Study of Urdu Version of Knee Outcome Survey-Activities of Daily Living Scale
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00298
Record Dates: First submitted 2022-02-01; First posted 2022-02-02 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Knee Pain
Keywords: Knee Outcome Survey-Activities of Daily Living Scale; General Population; Cultural adaptation; Validity; Urdu Version; Reliability; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to translate Knee Outcome Survey-Activities of Daily Living Scale into Urdu language and to check the reliability and validity of the Knee Outcome Survey-Activities of Daily Living Scale in Urdu language for the general population of Pakistan

DETAILED DESCRIPTION:
Approximately 150 participants will be included in the study on the basis of inclusion and exclusion criteria. The English version of the Knee Outcome Survey-Activities of Daily Living Scale will be translated and culturally adapted as per as previous recommendations. In the general population with knee pain,Urdu version of the Knee Outcome Survey-Activities of Daily Living Scale will be distributed among general participants by choosing convenience sampling technique based on predefined inclusion and exclusion criteria. To test inter and intra-observer reliability of the final Urdu version of Knee Outcome Survey-Activities of Daily Living Scale with Knee osteoarthritis outcome survey and Lysholm knee score will be filled within same day, by two observers and for the inter-observers assessment, with an interval of 30 minutes between the first and second application. Third assessment will carry out after 7 days by Observer-1(re-intra-observers assessment. Data will be entered and analyzed by Cronbach alpha value.Test-retest reliability will be assessed using interclass correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* Ability to walk without assistive device
* proficiency in the Urdu language
* pain level of at least 30% on the visual analog scale

Exclusion Criteria:

* Other osteoarthropathies with a good history
* If you have a heart condition or are having trouble with your nerves
* A debilitating factor that lowers functional independence and activity levels
* A lower-extremity fracture within the previous six months of the research
* Other joint diseases include ligament, menisci, or patellofemoral issues, as well as severe non-osteoarthritic knee effusion or arthroplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pakistani population with knee osteoarthritis was included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Knee outcome survey-Activities of daily living scale | 1st day
  Its purpose is to assess the knee's functional state in relation to disability and disease It is a self-reported tool for individuals with knee osteoarthritis. The Knee Outcome Survey is divided into two scales. We may use the Activities of Daily Living Scale to evaluate symptoms and limitations in daily living functions
Knee osteoarthritis outcome scale | 1st day
  The Knee osteoarthritis outcome scale evaluates both the short- and long-term effects of knee injuries. Pain, other Symptoms, Function in Daily Living, Function in Sport and Recreation, and knee-related Quality of Life are among the 42 questions in five independently scored sub-scales.
Lysholm knee scoring scale | 1st day
  The Lysholm knee scale has eight domains: limping, locking, pain, stair-climbing, support, instability, swelling, and squatting.A total score of 0 to 100 is generated, with 95 indicating an outstanding outcome, 84 suggesting a good result, 65 indicating a fair result, and 65 indicating a bad result. The Lysholm knee scale has been used to assess a wide range of knee problems.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No